CLINICAL TRIAL: NCT01778881
Title: Effectiveness of Physical Therapy Interventions, Relative to Dental Treatment in Individuals With Bruxism: a Randomized Clinical Trial
Brief Title: Physical Therapy Interventions Relative to Dental Treatment in Individuals With Bruxism
Acronym: Bruxism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cinthiamiotto
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-06

CONDITIONS: Bruxism
Keywords: Bruxism; Physical therapy modalities; Massage; Muscle stretching exercises; Relaxation therapy; Imagination
MeSH Terms: conditions — Bruxism | interventions — Massage; Dental Care; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Massage + Exercise (Experimental): Massage and stretching exercises
  Interventions: Other: Massage and stretching exercises
- Relaxation +Imagination (Experimental): Relaxation and Imagination therapies
  Interventions: Other: Relaxation and imagination therapies
- Dental treatment (Experimental): Reconstruction with composite resin
  Interventions: Other: Dental treatment
- Massage + Exercise + Relaxation + Imagination (Experimental): Massage, stretching exercises, relaxation and imagination
  Interventions: Other: Massage, exercises, relaxation and imagination therapies

INTERVENTIONS:
Other: Massage and stretching exercises — The routine to be used in this group (stretching, massage, and diaphragmatic breathing).
  Arms: Massage + Exercise
Other: Relaxation and imagination therapies — The routines to be adopted will focus on progressive muscle relaxation associated to imagination and diaphragmatic breathing.
  Arms: Relaxation +Imagination
Other: Dental treatment — Restoring treatment will involve direct reconstruction of the anterior guides (incisive faces of the incisive and canine teeth) with resin.
  Arms: Dental treatment
Other: Massage, exercises, relaxation and imagination therapies — The routine to be used in this group (stretching, massage, diaphragmatic breathing, progressive muscle relaxation and imagination therapies).
  Arms: Massage + Exercise + Relaxation + Imagination

SUMMARY:
Bruxism is a parafunctional habit characterized by grinding and/or clenching of the teeth. It may happen while awake (awake bruxism) or while sleeping (sleep bruxism). In adults, the prevalence is 20% for the awake bruxism and 8% for the sleep bruxism. Peripheral, central, and psychosocial factors influence the disorder, which may predispose to pain in the masticatory muscles and neck, headache, decreased pain thresholds in the masticatory and cervical muscles, limitation mandibular opening, sleep disorders, stress, anxiety, depression, and overall impairment of oral health. The aim of this study is to compare physical therapy interventions with dental treatment in pain, mandibular opening, sleep quality, anxiety, stress, depression, and oral health in individuals with bruxism.

DETAILED DESCRIPTION:
Participants will be randomized into one of four groups: Group 1 (n = 24) intervention will consist of massage and stretching exercises; Group 2 (n = 24) will consist of relaxation and imagination therapies; Group 3 (n = 24) will receive dental treatment and Group 4 (n=24) will consist of massage, exercises, relaxation and imagination. The evaluations will be performed at baseline, immediately after treatment, and at 2-month follow-up. Pain intensity will be assessed using the visual analogical scale, while pain thresholds will be determined using algometry. Mandibular opening will be assessed using digital pachymeter. Sleep quality will be assessed by the Pittsburgh Sleep Quality Index, anxiety by the State-Trait Anxiety Inventory, stress by the Perceived Stress Scale-10, depression by the Beck Depression Inventory, and oral health will be assessed using the Oral Health Impact Profile - 14. Significance level will be determined at the 5% level.

Valid Reasons of updates:

2014 - Changes made according requeriments of plattform of ClinicalTrials.

2015 - In 2014, in my qualification examination at University of São Paulo, the professors suggested my transfer from master degree to direct doctorate and the inclusion of more one intervention group, whereas the other three groups were still in the randomization process. I updated the registration in 2015 with the inclusion of this fourth group. However, as the protocol published in 2014 reports 3 groups (initial idea of the master degree before the transition to the direct doctorate), this fourth group started the treatment (massage, exercises, relaxation and imagination) after the end of treatment of other three groups (Groups:1,2 and 3).

2016- Although I have listed as primary variables: pain (VAS) and mandibular opening in this platform in 2013, and in the protocol published in 2014 (http://trialsjournal.biomedcentral.com/articles/10.1186/1745-6215-15 -8); symptoms like clenching, headaches and sleep difficulties were also assessed by VAS, and no included posteriorly to trial registration. They were evaluated, but not described in this platform. The same happened with intention to treat analysis.

June 20, 2016- Updates for clarifications and suggested by the PRS Team.

Please, any doubts, send me a e-mail! Thank you!

ELIGIBILITY:
Inclusion Criteria:

* Sleep Bruxism identified by the interview, clinical assessment and diagnostic criteria of the International Classification for Sleep Disorders (ICSD) of the American Academy of Sleep Medicine (AASM);
* Awake bruxism identified by the interview, clinical assessment and questionnaire of Pintado;
* Aged between 18 to 60 years;
* A minimum pain intensity score of 3 on the Visual Analogical Scale.

Exclusion Criteria:

* More than two missing teeth, except third molars;
* Systemic and/or degenerative diseases;
* Arthrogenic or mixed temporomandibular disorder (TMD) according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD), axis I;
* Neurological or psychiatric diseases (with the exception of anxiety and depression);
* Using medications that influence sleep or motor behavior;
* Periodontal disorders;
* Abuse of alcohol and/or illicit drugs;
* Removable dentures, superior and/or inferior;
* Total dentures;
* Direct trauma or past surgery in the orofacial region;
* On physical, speech, dental, or psychological therapy at the time of study entry.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain / Mandibular opening | 6 weeks
  Visual Analogical Scale (VAS), pain thresholds (algometry) and mandibular opening (digital pachymeter)

SECONDARY OUTCOMES:
Sleep Quality | 6 weeks
  Pittsburgh Sleep Quality Index (PSQI)
Anxiety | 6 weeks
  State-Trait Anxiety Inventory (STAI)
Stress | 6 weeks
  Perceived Stress Scale (PSS)
Depression | 6 weeks
  Beck Depression Inventory (BDI)
Oral Health Quality | 6 weeks
  Oral Health Impact Profile (OHIP-14)

CONTACTS AND LOCATIONS:
Overall Officials: Amélia P Marques, PhD, Study Director — University of Sao Paulo; Cinthia SM Amorim, MSc, Principal Investigator — University of Sao Paulo
Locations (1):
- Medicine School of the University Of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santos Miotto Amorim C, Firsoff EF, Vieira GF, Costa JR, Marques AP. Effectiveness of two physical therapy interventions, relative to dental treatment in individuals with bruxism: study protocol of a randomized clinical trial. Trials. 2014 Jan 7;15:8. doi: 10.1186/1745-6215-15-8. PMID 24398115